CLINICAL TRIAL: NCT00459641
Title: A Phase 2 Randomised, Open-label, Multi-centre Ascending Dose Study of the Efficacy, Safety and Tolerability of I-040302 Versus Control Injection (Bone Marrow Aspirate or Steroids) in Children and Young Adults With Solitary Bone Cysts
Brief Title: Safety and Tolerability of I-040302 in Children and Young Adults With Solitary Bone Cysts
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Stopped before any site initiation or any recruitment due to change in overall product development plan
Sponsor: Kuros Biosurgery AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS I-040302/01
Record Dates: First submitted 2007-04-11; First posted 2007-04-12 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Bone Cysts
Keywords: Osteogenic Gel; Solitary Bone Cysts
MeSH Terms: conditions — Bone Cysts | interventions — Standard of Care; Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): I-040302 doses of up to 1 mg, 2 mg or 4 mg of TGplPTH1-34
  Interventions: Drug: I-040302
- 2 (Active Comparator): Standard of care (bone marrow aspirate or steroids)
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: I-040302 — doses of up to 1 mg, 2 mg or 4 mg of TGplPTH1-34
  Arms: 1
Other: Standard of Care — Bone marrow aspirate or steroids
  Other Names: Bone marrow aspirate or steroids
  Arms: 2

SUMMARY:
This is a randomised, controlled, open-label study of a single intralesional administration of I-040302 or a single bone marrow aspirate or a single steroid injection (methylprednisolone). Subjects will undergo screening with X-ray and magnetic resonance imaging (MRI) in the diagnosis of a solitary bone cyst.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 6 - 16 years of age
2. Diagnostic evidence of unicameral bone cysts based on one or more of a combination of any of the following methods:

   * Cyst fluid examination
   * Plain radiographs
   * MRI
3. Subjects with the following types of cysts:

   * Intact cysts that are either growing or at risk of fracture, requiring surgical intervention
   * Persistence of a cyst cavity following cyst fracture that has received conservative treatment/s to repair the fracture
   * Persistence of a cyst cavity despite repeated interventions
4. Subjects with bone cyst volumes < 30 mL
5. Subjects must be appropriately communicative to verbalise pain.
6. Subjects must be able to understand and be willing to comply with the protocol procedures.
7. Subjects who have provided written informed consent to participate in the study
8. The legally authorised representative of the child must give written informed consent after the child has agreed to participate in the study.

Exclusion Criteria:

1. A history of/or presence of active cancer
2. Family history of retinoblastoma
3. Indication of aneurysmal bone cyst on MRI, cyst aspiration or histology
4. Possible presence of osteosarcoma or uncertain histology
5. Systemic or localised infection at time of surgery
6. Evidence of immune-suppression
7. Evidence of hypercalcemia
8. Cyst volume > 30 mL
9. Fracture present in the cortical bone surrounding the cyst
10. Evidence of rapid venous drainage from the cyst determined by rapid disappearance of X-ray contrast medium during the surgical process.
11. Suspected or known evidence of allergic reactions towards any of the components of I-040302
12. Known clinically significant organ or systemic diseases such that, in the opinion of the investigator, the significance of the disease will compromise the subject's participation in the study
13. Pregnant or lactating females
14. Participation in another clinical trial within 3 months prior to trial start

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2014-06 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Radiographic images | At 6 months and throughout the study

SECONDARY OUTCOMES:
Blood parameters | At 6 months and throughout the study
Vital signs | At 6 months and throughout the study
Questionnaires of life questionnaire | At 6 months and throughout the study
Pharmacoeconomic evaluation | At 6 months and throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Jamieson, MD, Study Director — Kuros Biosurgery AG, Technoparkstrasse 1, CH-8005 Zurich